CLINICAL TRIAL: NCT02309788
Title: Radiotherapy in Hepatocellular Carcinomas After Hepatectomy With Narrow Margin (<1 cm) or Portal Vein Thrombosis
Acronym: RHCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, TaoBai, Researcher, Guangxi Medical University
Other Study IDs: TAOBAI
Record Dates: First submitted 2014-12-02; First posted 2014-12-05 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: HepatoCellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- RT: Resectable HCC patients adjuvant RT for PVT or NM
- No RT: Resectable HCC patients adjuvant other treatment for PVT or NM

SUMMARY:
Hepatocellular carcinoma (HCC) is one of ten leading cancer types worldwide and also in Asia, but the five-year relative survival rate is relatively quite low1-3. As a common complication of HCC, portal vein tumor thrombosis (PVTT) have been reported with an occurrence of 34% ~ 50% in advanced HCC and it is now become an extremely pressing problem for hepatic surgeon. Nevertheless, the patients overall survival (OS) varies on their clinical features or liver function4. For HCC PVTT treatment, current options are surgical resection, embolization chemotherapy, radiation therapy, a variety of ablation therapy, biological and gene therapy,etc. Among them, the use of radiation therapy is getting more and more attention, and it is changing from the past palliative treatment to current curable treatment. From an oncologic point of view, a narrow margin <1 cm is not safe and is often associated with higher rates of recurrence and shorter patient survival.On the other hand, it is also believed that most intrahepatic recurrences arise from multicentric carcinogenesis and are distant from the resection margin.To address this issue, the investigators are going to conduct a series of retrospective and prospective studies to investigate the effect of adjuvant RT for centrally located HCC after narrow margin (<1 cm) hepatectomy on tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* HCC with no preoperative RT
* resectable lesion that could be completely removed, at the same time retaining a sufficient residual liver tissue to maintain adequate function
* compensated cirrhosis or no cirrhosis; Child-Pugh A
* ECOG Performance Status of 0 or 1.
* Patients who had undergone transarterial chemoembolization (TACE) were eligible for enrollment in the study, provided this form of therapy ended at least 4 weeks before study entry

Exclusion Criteria:

* unresectable hepatocellular carcinoma patients
* Hepatocellular carcinoma without portal vein tumor thrombus
* Hepatectomy without narrow margin(more than 1cm)
* presence of distant metastasis
* palliative resection with tumor residual
* non-HCC confirmed by postoperative pathology

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with HCC at the Affiliated Tumor Hospital of Guangxi Medical University Science were considered for enrollment in the study. The diagnostic criteria for HCC used in the study were in accordance with the American Association for the Study of Liver Diseases' 2005 guidelines. All patients had preoperative serum a-fetoprotein (AFP) levels >200 ng/mL or a typical enhancement pattern (arterial enhancement and portal/delayed washed out) on dynamic imaging of hepatic mass(es)>2 cm, or cytologic/histologic evidence of HCC
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- TaoBai, Nanning, Guangxi, China